CLINICAL TRIAL: NCT05141227
Title: Two-stage Open Reduction and Internal Fixation Versus Single-stage External Fixation for Complex Intra-articular Distal Tibial Fractures : A Randomized Controlled Trial
Brief Title: Two-stage ORIF Vs Ex. Fix. in Complex Pilon Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Osama Mohamed Eissa, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Complex pilon fractures
Record Dates: First submitted 2021-10-07; First posted 2021-12-02 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Pilon Fracture
MeSH Terms: interventions — Fracture Fixation, Internal

STUDY DESIGN:
Intervention Model Description: Open reduction and internal fixation versus external fixation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- two stage ORIF (Experimental): Two-stage Open reduction and internal fixation
  Interventions: Procedure: Two-stage Open reduction and internal fixation ( ORIF) using plates & screws
- single stage Ex. Fix (Experimental): Single-stage external fixation with minimal internal fixation if needed
  Interventions: Procedure: single-stage external fixation (EX.FIX.) with minimal internal fixation using cannulated screws if needed

INTERVENTIONS:
Procedure: Two-stage Open reduction and internal fixation ( ORIF) using plates & screws — Two stage ORIF using initially temporary spanning fixator then conversion to plates & screws
  Arms: two stage ORIF
Procedure: single-stage external fixation (EX.FIX.) with minimal internal fixation using cannulated screws if needed — Single stage Ex.Fix. Using illizarov & minimal fixation of the articular surface using cannulated screws through mini open approaches
  Arms: single stage Ex. Fix

SUMMARY:
This study aims to compare the clinical, radiological, and functional outcomes of two-stage open reduction and internal fixation with single-stage external fixation in the treatment of comminuted tibial pilon fractures.

DETAILED DESCRIPTION:
A pilon fracture ( also known as tibial plafond fractures) is a fracture of the distal end of the tibia with comminution, intra-articular extension and significant soft tissue injury.Pilon injury accounts for about 5% to 10% of all tibial fractures, and for <10% of lower extremity injuries. The incidence rate is relatively low. However, with the high incidence of high energy trauma and accidental falls, the number of comminuted fractures has increased in recent years.Among all pilon fractures, about 30% are complex pilon fractures (AO/ OTA 43C type) caused by high-energy injuries.

Most complex pilon fractures are associated with severe soft tissue injuries, making the treatment challenging. Optimal treatment of comminuted pilon fractures requires precise anatomical reduction accompanied by early functional exercise. Several methods have been advocated to manage complex pilon fractures, but an optimal fixation technique remains controversial.

In 1979, Ruedi and Allgower first reported satisfactory results with primary open reduction and internal fixation.However, many authors have noted significant complications when open reduction and internal fixation was applied to severe pilon fractures, including an infection rate as high as 55%, wound necrosis and skin sloughing. These complications arose from the internal fixation, leading many orthopaedic surgeons to choose external fixation as an alternative.

Although external fixation decreased wound necrosis and skin sloughing, high rates of pin site infection and malalignment with subsequent non-union occurred. Therefore, orthopaedic surgeons made great efforts to establish methods that provided good results and decreased postoperative complications.

With the accumulation of surgical experience and the development of surgical techniques, two-stage open reduction and internal fixation and limited internal fixation combined with external fixation were established, and these two methods are now widely advocated for the treatment of comminuted tibial pilon fractures.

Two-stage open reduction and internal fixation involves closed reduction and external fixation followed by conversion to open reduction and internal fixation after the condition of the surrounding soft tissues has improved. This technique focuses on the soft tissue condition and potentially decreases the incidence of soft tissue complications.Thus, this method is widely considered the standard of care for high-energy pilon fractures.

However, other surgeons have recommended limited internal fixation combined with external fixation for these severe fractures as an alternative to open reduction and internal fixation to reduce the risk of postoperative complications.

The CT based four-column classification has been adopted by many surgeons as a guide for the treatment of comminuted pilon fractures.

The four-column classification can be summarized as lateral column (the distal fibula), posterior column (the posterior part of the intermalleolar line with the distal tibial shaft), anterior column (the anterior part of the intermalleolar line with the distal tibial shaft) and medial column (the medial one-third of the tibial plafond with the distal tibial shaft) Till now, there's no randomized prospective controlled trials confirmed which method either two-stage open reduction and internal fixation or single-stage external fixation is superior regarding clinical, radiological, and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients
* Both males and females
* Closed or open (grade 1&2) pilon fractures according to Gustilo and Anderson classification
* AO/OTA type C fractures
* Compromised soft tissue not allowing for primary open reduction and internal fixation
* Unilateral or bilateral
* Isolated or polytrauma patients

Exclusion Criteria:

* Skeletally immature patients
* Open grade 3 pilon fractures
* Patients eligible for primary open reduction and internal fixation
* Ipsilateral lower limb fractures
* Pathological fractures
* Pre-existing symptomatic ankle arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Functional | 12 months
  Functional outcome will be assessed using the American Orthopaedic Foot and Ankle Society (AOFAS) evaluation system.
  The score includes I.Pain (40 point) II. Function (50 points) It's divided into 7 items
  1. Activity limitations, support requirements (10points)
  2. Maximum walking distance, blocks (5 points)
  3. Walking surfaces (5 points)
  4. Gait abnormality (8 points)
  5. Sagittal motion (flexion plus extension) (8points)
  6. Hindfoot motion (inversion plus eversion) (6points)
  7. Ankle-hindfoot stability (anteroposterior, varus-valgus) (8 points) III. Alignment(10 points) IV. Total Score(100 points)
Radiological | 12 months
  Accuracy of reduction in plain x Ray using burwell& charnely score It includes Anatomical reduction , fair reduction & poor reduction
  1. Anatomical...
     * No medial or lateral displacement of the medial & lateral malleulus
     * no angulation
     * no more than 1 ml of longitudinal displacement of the medial or lateral malleli
     * no more then 2 ml of proximal displacement of a large posterior fragment
     * no talus displacement
  2. Fair ...
     * No medial or lateral displacement of the medial & lateral malleulus
     * no angulation
     * 2-5 ml of posterior displacement of lateral malleulus
     * 2-5 ml of proximal displacement of a large posterior fragment
     * no talus displacement
  3. Poor ...
     * Any medial or lateral displacement of the medial & lateral malleulus
     * no angulation
     * more than 5 ml of posterior displacement of lateral malleulus
     * more than 5 ml of proximal displacement of a large posterior fragment
     * any residual talus displacement

CONTACTS AND LOCATIONS:
Overall Officials: Salah Abou-Seif, Professor, Study Chair — Faculty of medicine, Ain Shams University
Locations (1):
- El-Demerdash hospital Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mauffrey C, Vasario G, Battiston B, Lewis C, Beazley J, Seligson D. Tibial pilon fractures: a review of incidence, diagnosis, treatment, and complications. Acta Orthop Belg. 2011 Aug;77(4):432-40. PMID 21954749
- [Background] Ruedi TP, Allgower M. The operative treatment of intra-articular fractures of the lower end of the tibia. Clin Orthop Relat Res. 1979 Jan-Feb;(138):105-10. PMID 376196
- [Result] Michelson J, Moskovitz P, Labropoulos P. The nomenclature for intra-articular vertical impact fractures of the tibial plafond: pilon versus pylon. Foot Ankle Int. 2004 Mar;25(3):149-50. doi: 10.1177/107110070402500307. PMID 15006336
- [Derived] Eissa MO, Thakeb MF, AbouSeif S, Fayyad TA, Alkersh MA, ElGebeily MA, Aly AS, Baraka MM. Comparison of two-stage open reduction and internal fixation and single-stage external fixation for complex pilon fractures: a randomized controlled trial. Int Orthop. 2025 Nov 13. doi: 10.1007/s00264-025-06682-2. Online ahead of print. PMID 41225168